CLINICAL TRIAL: NCT06746103
Title: RELIEVE Research on Effectiveness of Surgery and Radiotherapy on Relieving Spine Tumor Pain in Patients with Vertebral Metastases
Brief Title: RELIEVE: Research on Effectiveness of Surgery and Radiotherapy on Relieving Spine Tumor Pain in Patients with Vertebral Metastases
Acronym: RELIEVE
Status: Not yet recruiting | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: RELIEVE
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Spinal Metastasis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgery — Surgery may be instrumented stabilization surgery alone, instrumented stabilization and decompression, or decompression surgery alone.

SUMMARY:
This is a prospective, multicenter, observational study focusing on assessing and managing pain in patients with metastatic spinal tumors. Pain from spinal metastases adversely impacts quality of life, function, and treatment outcomes. Advances in surgical techniques have shown significant benefits. However, previous studies either lacked nuanced differentiations or simply categorized pain as mechanical or non-mechanical; explaining the highly variable pain outcome measurements in these studies. This study employs the AO Spine Cancer-Related Pain Classification to better categorize neoplastic spinal pain by etiology.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational study. Patients with metastatic spinal tumors and one symptomatic metastatic site (ie, the index metastasis) that is causing at least one type of pain (ie, the index pain) of interest to this study that has at least "moderate" pain in intensity (numeric rating scale [NRS] > 4) will be enrolled from participating sites. Four types of neoplastic pain in the AO Spine Cancer-Related Pain Classification are of interest to this study.

1. The axial non-triggered pain is hypothesized to be secondary to periosteal stretching and/or release of nociceptive cytokines; it is mostly associated with osteoclastic activity but can be sometimes associated with reactive sclerosis. This pain may show a diurnal variation with increased severity at night and typically responds to steroids or opioid medications.
2. The axial triggered/mechanical pain is nociceptive pain secondary to inability of osseous spinal structures to support physical loads. It is typically associated with osteoclastic activity but can also be due to periosteal nerve stimulation from frank fractures or microfractures. This pain typically does not respond well to the medical treatments and if the pain is severe, progressive, or debilitating, may benefit from stabilization.
3. Radicular non-triggered pain is a result of persistent compression of a nerve root which can be due to tumor or bone expansion. This type of neurologic pain follows a specific nerve root distribution with a correlative compression lesion. It may be resolved with decompression or potentially with nonoperative measures such as radiotherapy or systemic treatments.
4. Radicular triggered/mechanical pain is a result of transient compression of a nerve root caused by mechanical instability. This type of neurologic pain also follows a specific nerve root distribution with a correlative compression lesion. It may be relieved in certain position such as recumbency and often benefits from stabilization surgery with or without decompression.

Patients will be treated (ie, the index treatment) with surgery alone, surgery with postoperative radiotherapy, or radiotherapy alone for the index metastasis. Day 0 is defined as: 1) for patients receiving surgery only, the day of the surgery (or the first stage of surgery in the case of staged surgery), 2) for patients receiving radiotherapy only, the day of the first session of radiotherapy, or 3) for patients receiving both surgery and radiotherapy, whichever treatment day that comes earlier. Patients will be followed up at 1 month, 3 months, and 6 months after Day 0. The primary study outcome is the intensity of the four different types of pain caused by the index spinal metastasis. The study will delineate how these kinds of pain respond to treatment over time. Secondary objectives investigate factors predictive of pain relief and the relationship between pain and other patient-reported outcomes (PROs).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients diagnosed with metastatic spinal tumors with one index metastatic site that, confirmed by the treating clinicians, is causing spine pain
* Patients experience at least one type of pain that is of interest of this study, namely, axial non-triggered pain, axial triggered/mechanical pain, radicular non-triggered pain, and radicular triggered/mechanical pain
* At least one type of the pain experienced has an NRS > 4 of 10
* Patients undergoing surgery and/or radiotherapy

  * Surgery may be instrumented stabilization surgery alone, instrumented stabilization and decompression, or decompression surgery alone.
  * Percutaneous screw fixation counts as instrumented stabilization surgery.
  * Any kind of radiotherapy is includable.
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Estimated survival < 3 months
* Patients with more than one symptomatic spine metastasis site

  o An example is a patient with two metastasis sites: a lumbar metastasis (causing vertebral fracture and epidural compression leading to mechanical lower back pain and static radicular pain to legs) and a cervical metastasis (causing tumor-related pain at the neck).
* Patients with other sources of pain that may confound the measurement of the primary outcome

  o An example is a patient with liver metastasis which causes visceral pain that can confound the thoracic spinal pain caused by the spinal metastasis.
* Patients undergoing the following treatments alone without the surgeries listed in the inclusion criteria or radiotherapy

  * Cement augmentation, vertebroplasty, kyphoplasty, and other emerging interventions such as local ablative technique
  * Chemotherapy or systemic therapy alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic spinal tumors as per eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity on the Brief Pain Inventory Intensity Scale of four different types of pain caused by the index spinal metastasis, measuring pain on a numeric rating scale from 0 to 10, with 0 meaning no pain and 10 meaning as bad as one can imagine. | Baseline and 3 months
  The primary study outcome is the intensity of the four different types of pain caused by the index spinal metastasis, ie, the index pain(s):
  * Axial non-triggered pain
  * Axial triggered/mechanical pain
  * Radicular non-triggered pain
  * Radicular triggered/mechanical pain

SECONDARY OUTCOMES:
Patient Reported Outcome Measure: Michigan Body Map measuring pain location | Baseline, 1 month, 3 months, and 6 months
  The following Patient Reported Outcome Measure will be measured: Michigan body map. The Michigan Body Map is used to record the location and number of painful body regions. At baseline, patients will use the map to indicate the locations of each index pain experienced. At 1 month, 3 months, and 6 months, patients will use the map to indicate any new locations of pain, apart from the locations of the index pain, since the index treatment.
Patient Reported Outcome Measure: PainDETECT measuring neuropathic pain | Baseline, 1 month, 3 months, and 6 months.
  The following Patient Reported Outcome Measure will be measured: PainDETECT Questionnaire. The PainDETECT Questionnaire was initially developed as a screening tool to detect neuropathic pain component in patients with chronic low back pain. The questionnaire consists of seven items describing neuropathic pain symptoms, with item responses ranging from 0 (never) to 5 (very strongly), as well as one item each describing temporal pain patterns (four patterns with scores ranging from -1 to +1) and presence of radiating pain (if yes, score of +2). The total score ranges from 0 to 38, with higher score indicating higher likelihood of a neuropathic pain component.
  Patients will fill in the PainDETECT Questionnaire at baseline, 1 month, 3 months, and 6 months.
Patient Reported Outcome Measure: BAT measuring breakthrough pain | Baseline, 1 month, 3 months, and 6 months.
  The following Patient Reported Outcome Measure will be measured: Breakthrough Pain Assessment Tool (BAT). Breakthrough pain is defined as "a transient exacerbation of pain that occurs either spontaneously, or in relation to a specific predictable or unpredictable trigger, despite relatively stable and adequately controlled background pain".
  The BAT questionnaire comprises 14 items, including nine related to pain and five related to its management. The first question uses body shape to locate the painful areas. The remaining items include free text (four questions), 10-point rating scale (six questions), and categorical scale (three questions).
  Patients will fill in the BAT at baseline, 1 month, 3 months, and 6 months.
Patient Reported Outcome Measure: PROMIS Bank v1.0-Fatigue measuring fatigue | Baseline, 1 month, 3 months, and 6 months.
  The following Patient Reported Outcome Measure will be measured: PROMIS Bank v1.0-Fatigue. The PROMIS Bank v1.0-Fatigue instrument will be used to assess fatigue and fatigue interference in the past 7 days. The item responses are Likert-scale responses ranging from 1 (never) to 5 (always) with higher scores indicating greater fatigue or fatigue interference.
  Patients will complete the PROMIS Bank v1.0-Fatigue instrument at baseline, 1 month, 3 months, and 6 months.
Patient Reported Outcome Measure: PROMIS Bank v2.0-Physical Function measuring physical function | Baseline, 1 month, 3 months, and 6 months.
  The following Patient Reported Outcome Measure will be measured: PROMIS Bank v2.0-Physical Function. The PROMIS Bank v2.0-Physical Function instrument will be used to assess physical function. The item responses are Likert-scale responses ranging from 1 (unable to do/cannot do/cannot do because of health/not at all) to 5 (without any difficulty/not at all/no difficulty at all/completely) with higher scores indicating better physical function.
  Patients will complete the PROMIS Bank v2.0-Physical Function instrument at baseline, 1 month, 3 months, and 6 months.
Patient Reported Outcome Measure: RAPA measuring physical activity | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: Rapid Assessment of Physical Activity (RAPA). The RAPA instrument will be used to assess patients' physical activity levels. It consists of nine items with item responses of yes and no. The RAPA instrument categorizes the individuals into five categories of physical activity: sedentary, under-active, under-active regular-light activities, under-active regular, and active.
  Patients will complete the RAPA instrument at baseline and 3 months.
Patient Reported Outcome Measure: SOSGOQ v2 measuring health-related quality of life | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: The Spine Oncology Study Group Outcomes Questionnaire, version 2 (SOSGOQ v2). The SOSGOQ v2 will be used to assess patients' health-related quality of life. It is a questionnaire developed specifically for patients with metastatic spine disease. The SOSGOQ contains 20 items representing all four domains of the International Classification of Function and Disability. Additionally, there are seven FU questions referring to treatment satisfaction. It is made up of five domains: physical function, neural function, pain, mental health, and social function.
  Patients will complete the SOSGOQ v2 at baseline and 3 months.
Patient Reported Outcome Measure: GAD-7 measuring anxiety | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: General Anxiety Disorder-7 (GAD-7). The GAD-7 questionnaire will be used to screen for generalized anxiety disorders. It consists of seven items about how often the patient experiences each item over the past 2 weeks, with item responses ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher score indicating greater level of anxiety. A total score of 15-21 is considered severe anxiety.
  Patients will complete the GAD-7 questionnaire at baseline and 3 months.
Patient Reported Outcome Measure: PHQ-8 measuring depression | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: Patient Health Questionnaire-8 (PHQ-8). The PHQ-8 questionnaire will be used to assess depression. It consists of eight items about patients' experiences in the past 2 weeks, with item responses ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 24, with higher score indicating more distress. A score of 10 or greater is considered major depression, and 20 or more is severe major depression.
  Patients will complete the PHQ-8 questionnaire at baseline and 3 months.
Patient Reported Outcome Measure: PROMIS Bank v1.0-Sleep Disturbance measuring sleep | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: PROMIS Bank v1.0-Sleep Disturbance. The PROMIS Bank v1.0-Sleep Disturbance instrument will be used to assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep in the past 7 days. The item responses are Likert-scale responses ranging from 1 (always/very good) to 5 (never/very poor) with higher scores indicating more sleep disturbance.
  In addition, sleep duration will be assessed as the average number of hours and minutes of actual sleep obtained per night during the past month.
  Patients will complete the PROMIS Bank v1.0-Sleep Disturbance instrument and the question on sleep duration at baseline and 3 months.
Patient Reported Outcome Measure: PCS -6 measuring pain catastrophizing | Baseline and 3 months.
  The following Patient Reported Outcome Measure will be measured: The Pain Catastrophizing Scale-6 (PCS-6). The PCS-6 comprises 6 items assessing catastrophic thoughts or feelings accompanying the pain experience, with item responses ranging from 0 (not at all) to 4 (all the time). The total score of PCS-6 ranges from 0 to 24.
  Patients will complete the PCS-6 at baseline and 3 months.
Patient Reported Outcome Measure: PEPSO measuring patient expectations | Baseline.
  The following Patient Reported Outcome Measure will be measured: The Patient Expectations in Spine Oncology questionnaire (PEPSO). PEPSO evaluates patient expectation related to surgery and/or radiotherapy for symptomatic spinal metastases. The questionnaire has two versions (surgery versus radiotherapy). There are 13 items regarding expected outcomes, 3 items regarding prognosis and 6 items regarding consultation with spine surgeon/radiation oncologists. In this study, only English-speaking patients will complete the PEPSO questionnaire at baseline. For patients undergoing surgery followed by radiotherapy, the PEPSO questionnaire version for patients waiting for surgery will be used.
Patient Reported Outcome Measure: PGIC scale measuring global improvement with treatment | 1 month, 3 months, and 6 months.
  The following Patient Reported Outcome Measure will be measured: Patient's Global Impression of Change (PGIC) scale. The PGIC scale is recommended for use in chronic pain clinical trials as a core outcome measure of global improvement with treatment. The scale contains a single item with which the patients are asked to rate their improvement with treatment during a clinical trial on a 7-point scale with the options of "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," and "very much worse". Patients will complete the PGIC scale at 1 month, 3 months, and 6 months.
Time up and go test measuring mobility | Baseline, 1 month, 3 months and 6 months
  The following mobility test will be conducted to evaluate patients' mobility:
  - Time up and go test: measuring the time that the patient takes to rise from a chair, walks 3 meters, turn around 180 degrees, walks back to the chair, and sits down while turning 180 degrees.
30-second sit-to-stand test measuring mobility | Baseline, 1 month, 3 months and 6 months
  The following mobility test will be conducted to evaluate patients' mobility:
  - 30-second sit-to-stand test: measuring the number of stands completed within 30 seconds; more than halfway up at the end of 30 seconds counts as a full stand, and incorrectly executed stands are not counted.
6-minute walk test measuring mobility | Baseline, 1 month, 3 months and 6 months
  The following mobility test will be conducted to evaluate patients' mobility:
  - 6-minute walk test: measuring the distance in meters covered over 6 minutes.
Walking speed measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Walking speed (meters/second) measuring the time it takes to walk a specified distance.
Speed variability measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Speed variability, measuring the fluctuation in gait speed in meter/second.
Cadence measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Cadence measured by the number of steps/minute.
Step length measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Step length in centimeters: distance traversed during a step made with one leg, measured from the heel of the other leg to the heel of the measured leg
Stride length measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Stride length in centimeters, distance between two steps or initial contact of one foot to initial contact of same foot
Step length symmetry measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Difference between left and right step length, as a percentage of stride length
Single support measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Single support: percentage of time during a walk that one foot, and only that foot, is in contact with the ground
Stance measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Stance: percentage of time during a walk that one foot is in contact with the ground
Stance asymmetry measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Stance asymmetry: difference of time spent on right leg compared to left leg as a percentage of gait cycle
Double support measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Double support: percentage of time both feet are in contact with the ground
Double support asymmetry measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Double support asymmetry: percentage difference between the initial double support and the terminal double support
Step width measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Step width: width of a stride, as measured from heel to heel when both heels are in contact with the ground
Stride consistency measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Stride consistency: how similar strides are to one another within a walk, measured on a scale of 0 to 100, with 100 being a walk where each stride is exactly the same
Hip range of motion measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Hip range of motion: total range of motion for the hip in the sagittal plane during the gait cycle
Femoral rotation range measuring gait | Baseline, 1 month, 3 months and 6 months
  The following gait analysis will be conducted:
  - Femoral rotation range: combined amount of internal and external rotation of the hip and femur over the length of each stride
Survival | Baseline, 1 month, 3 months and 6 months
  Survival is measured by following up if the patient is still alive.
Tumor control | Baseline, 1 month, 3 months and 6 months
  Tumor control is measured for the primary spine tumor (improved, stable, progressing, not assessed) as well as metastatic spine tumor(s) (local control index lesion as well as non-index lesion, new metastatic site(s)/lesion(s) and activity of metastasis overall.

IPD SHARING:
Plan to Share IPD: Undecided